## Effect of Therapeutic Exercise on the Activation of the Neck Extensors in People With Chronic Neck Pain

INFORMED CONSENT (Last review date: 19 of September, 2016)

NCT02950909 ID: H1472552616890

## INFORMED CONSENT

Dear Mr./Mrs .:

This study aims to study the effect of different exercises on pain, disability and the activity of different cervical muscles. Your participation in it, apart from providing the possible benefits of the treatment, will be useful for future advances in the management of cervical pain.

We request your collaboration to:

- Completion of a series of questionnaires related to cervical pain and disability.
- Analysis of cervical range of motion and posture in sitting position.
- Measurement of pain threshold at cevical pressure using a pressure algometer.
- Measurement by surface and fine wire intramuscular electromyography of the cervical musculature.

The total estimated time for these measurements is 2 hours. These measurements will be taken at the beginning and at the end of the study. Treatment lasts for six weeks with a brief weekly review.

The risks of participating in the study are: slight pain, small bruising (rare) and infection (very rare) due to the insertion of the needle. The sterile conditions of the study and the performance by an expert neurophysiologist minimize these risks.

Your participation in this study is not mandatory, you can withdraw from participating in it at any time, without any justification and without this decision having any consequence.

If you participate, your personal data will be kept confidential throughout the study and after it, in strict compliance with Organic Law 15/1999, of December 13, on the Protection of Personal Data.

I have carefully read this Informed Consent, I have asked the physiotherapist responsible for my assessment all the doubts and questions that I have considered pertinent and I have been answered satisfactorily, for which I give my consent to be included in this study.

| Mr/Ms. : | | with DNI: |
|----------|-------|-----------|
| Date: | Sign: | |

## **INFORMED CONSENT TO USE THE IMAGE**

Universitat de València

| Mr/Ms: |
|---|
| With DNI |
| In accordance with the provisions of Organic Law 15/1999 on the Protection of Personal Data, I authorize that my image during the study may be used for scientific dissemination or for teaching at the university. |
| Signed: |
| First researcher: |
| Moisés Giménez Costa<br>Profesor asociado del Departamento de Fisioterapia<br>Facultad de Fisioterapia |